CLINICAL TRIAL: NCT02488980
Title: A Randomized, Double Blind, Placebo Controlled Evaluation of Weekly Tafenoquine (WR 238605/SB252263) Compared to Mefloquine for Chemosuppression of Plasmodium Falciparum in Western Kenya
Brief Title: An Evaluation of Weekly Tafenoquine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-9467
Record Dates: First submitted 2015-06-24; First posted 2015-07-02 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Falciparum Parasitaemia
Keywords: Falciparum Parasitaemia, Malaria
MeSH Terms: conditions — Malaria | interventions — tafenoquine; Mefloquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tafenoquine (Experimental): Tafenoquine 200 mg for three days followed by Tafenoquine 200 once a week for 24 weeks.
  Interventions: Drug: Tafenoquine
- Mefloquine (Active Comparator): Mefloquine 250 mg for three days followed by Mefloquine 250 once a week for 24 weeks.
  Interventions: Drug: Mefloquine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine 200 mg for three days followed by Tafenoquine 200 mg once a week for 24 weeks.
  Arms: Tafenoquine
Drug: Mefloquine — Mefloquine 250 mg for three days followed by Mefloquine 250 mg once a week for 24 weeks.
  Arms: Mefloquine
Drug: Placebo — Placebo for three days followed by placebo once a week for 24 weeks
  Arms: Placebo

SUMMARY:
This was a placebo controlled, randomised, double-blind, double-dummy study of the efficacy of weekly tafenoquine compared with weekly mefloquine or placebo in the chemosuppression of P. falciparum in Nyanza Province, western Kenya.

DETAILED DESCRIPTION:
Subjects were treated for 3 days with halofantrine to clear any existing parasitaemia. At the end of the clearance period, subjects free from malaria parasitaemia were randomized and received a loading dose of the study treatment (tafenoquine 200 mg, Mefloquine 250 mg or placebo) for tree days, followed by study treatment (tafenoquine 200 mg, mefloquine 250 mg or placebo, respectively) once a week for 24 weeks. After the treatment period subjects attended weekly follow-up safety visits until week 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers who provided informed consent (a healthy volunteer was defined as one who was free of ailments that might cause difficulty in evaluating drug efficacy or adverse experiences).
* Subjects aged 18-55 years.
* Subjects planning to reside in the study area for the entire study duration of approximately 70 weeks

Exclusion Criteria:

* Subjects with positive parasitaemia following halofantrine treatment for radical cure.
* Subjects with any medical condition which, in the opinion of the investigator, made the subject unsuitable to enter the study.
* Subjects with personal or family history of seizures.
* Female subjects with a positive serum beta-HCG5 (tested during screening and within 48 hours of first drug administration and approximately monthly thereafter).
* Women who were pregnant or lactating or who in the opinion of the investigator were at risk of becoming pregnant.
* Subjects with clinically significant abnormalities (to include but not limited to abnormal hepatic or renal function) as determined by history, physical and routine blood chemistries and haematology values. Subjects who had demonstrated hypersensitivity to any of the study drugs especially to any other 8-aminoquinolines.
* Subjects unwilling to report for drug administration or blood drawing during the 70 week duration of the study.
* Subjects with G6PD deficiency.
* Subjects with laboratory guideline values for exclusion: haemoglobin <10 gm/dL, platelets <80,000/mm3, WBC <3000ul3, creatinine or ALT more than twice the upper limit of normal for age.
* Subjects with an abnormal ECG, particularly an extended QTc interval > 0.42 seconds.
* Subjects taking any other anti-malarial product, or who had taken an antimalarial drug other than halofantrine within the previous two weeks.
* Subjects who had received an investigational drug (a new chemical entity not registered for use) within 30 days or 5 half-lives whichever was the longer.
* Subjects with a history of psychiatric disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2000-05; Primary Completion 2000-10 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Stoute, MD, Principal Investigator — Penn State Hershey Infectious Diseases

IPD SHARING:
Plan to Share IPD: Yes
SmithKline Beecham

REFERENCES:
- [Derived] Novitt-Moreno A, Ransom J, Dow G, Smith B, Read LT, Toovey S. Tafenoquine for malaria prophylaxis in adults: An integrated safety analysis. Travel Med Infect Dis. 2017 May-Jun;17:19-27. doi: 10.1016/j.tmaid.2017.05.008. Epub 2017 May 8. PMID 28495354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Kombewa Clinic, Kenya. 517 subjects were screened for entry in to the study. 211 of those subjects were not randomized to treatment due either to abnormal lab results, G6PD deficiency, extended QTc interval, failure to clear parasitaemia or "other" reason.
Period: Overall Study
Arm/Group | Tafenoquine | Mefloquine | Placebo
Started | 104 | 101 | 101
Completed | 102 | 99 | 99
Not Completed | 2 | 2 | 2
Not completed — Protocol Violation | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tafenoquine | Mefloquine | Total
Number analyzed (Participants) | 99 | 102 | 99 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 2 | 5
  Between 18 and 65 years | 98 | 100 | 97 | 295
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 33 | 105
  Male | 63 | 66 | 66 | 195
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 99 | 102 | 99 | 300
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 99 | 102 | 99 | 300

OUTCOME MEASURES:

1. Primary Outcome: Prophylactic Outcome Defined by the Subject Having no Positive Smears
Description: Prophylactic outcome (success/failure) at the end of the prophylactic treatment phase; outcome was based on absence/presence of asexual stage parasites of any Plasmodium species on a single blood smear.
Time Frame: 24 Weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Tafenoquine | Mefloquine
Number analyzed (Participants) | 99 | 102 | 99
participants
  Prophylactic Failure | 93 | 90 | 92
  Prophylactic Success (total) | 6 | 12 | 7
  Prophylactic Success (known) | 0 | 6 | 0
  Prophylactic Success (assumed) | 6 | 6 | 7

2. Secondary Outcome: Protective Efficacy Based on Two Consecutive Positive Smears
Description: Kaplan-Meier survival curves were produced for time to parasitaemia for both first positive smear and two consecutive positive smears. Analysis was based on a calculation of protective efficacy (PE) of tefaenoquine, defined as (1-relative risk of developing parasitaemia tafenoquine: placebo) x100% and 95.5% confidence intervals were constructed for the relative risk using Koopman's method.
Time Frame: 24 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Protective Efficacy
Arm/Group | Placebo | Tafenoquine | Mefloquine
Number analyzed (Participants) | 99 | 102 | 99
Percentage of Protective Efficacy | 0 [0 to 0] | 77.9 [59.7 to 88.2] | 56.8 [32.5 to 72.9]

3. Secondary Outcome: Time to a Single Positive Smear
Description: Kaplan-Meier survival curves were produced for time to parasitaemia for both first positive smear and two consecutive positive smears. 95.5% confidence intervals were constructed for the relative risk.
Time Frame: 24 Weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Tafenoquine | Mefloquine
Number analyzed (Participants) | 99 | 102 | 99
Days
  First positive smear | 43 [42 to 50] | 57 [53 to 70] | 50 [44 to 64]
  Two consecutive positve smears | 63 [57 to 79] | 0 [0 to 0] | 165 [154 to 165]

4. Other Pre Specified Outcome: Safety (SAEs and AEs)
Description: The most commonly reported experiences in subject occurring in at least 20% of subjects in any treatment group.
Time Frame: 28 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Tafenoquine | Mefloquine
Number analyzed (Participants) | 99 | 102 | 99
participants
  At least one AE | 92 | 98 | 97
  Headache | 37 | 45 | 49
  Upper Respiratory Tract Infection | 17 | 30 | 26
  Back Pain | 12 | 28 | 10
  Myalgia | 25 | 27 | 29
  Abdominal Pain | 24 | 25 | 19
  Coughing | 13 | 24 | 29
  Rhinitis | 21 | 12 | 20

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: Subjects with the most frequently reported AEs (>10 % of subjects in any treatment group)
Arm/Group | Placebo | Tafenoquine | Mefloquine
Serious Adverse Events (participants affected / at risk) | 4/101 | 10/104 | 2/101
Other Adverse Events (participants affected / at risk) | 92/101 | 98/104 | 97/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Tafenoquine (N=104) | Mefloquine (N=101)
Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) — Prophylaxis Treatment Period
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Prophylaxis Treatment Period
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Prophylaxis Treatment Period
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Prophylaxis Treatment Period
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Prophylaxis Treatment Period
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Prophylaxis Treatment Period
Unintended pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Prophylaxis Treatment Period
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Prophylaxis Treatment Period
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Prophylaxis Treatment Period
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) — Follow-up Period
Unintended pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Follow-up Period
Moniliasis GI (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Follow-up Period
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Follow-up Period
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Tafenoquine (N=104) | Mefloquine (N=101)
Headache (Nervous system disorders) | 37 (37) | 45 (45) | 49 (49)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 30 (30) | 26 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 28 (28) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (25) | 27 (27) | 29 (29)
Abdominal pain (Gastrointestinal disorders) | 24 (24) | 25 (25) | 19 (19)
Coughing (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 24 (24) | 29 (29)
Infection (Infections and infestations) | 20 (20) | 19 (19) | 14 (14)
Injury (Injury, poisoning and procedural complications) | 8 (8) | 18 (18) | 14 (14)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 14 (14) | 14 (14)
Gastroenteritis (Gastrointestinal disorders) | 9 (9) | 13 (13) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 13 (13) | 11 (11)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 12 (12) | 20 (20)
Dizziness (Nervous system disorders) | 7 (7) | 12 (12) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 12 (12) | 10 (10)
Conjunctivitis (Infections and infestations) | 13 (13) | 12 (12) | 7 (7)
Viral infection (Infections and infestations) | 7 (7) | 5 (5) | 11 (11)

LIMITATIONS AND CAVEATS:
Due to high failure rate a DMC was setup to assess if it was appropriate to continue study. DMC concluded that the study should continue in order to meet secondary objectives of evaluating the long-term safety and efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No